CLINICAL TRIAL: NCT00203411
Title: A Phase II Trial to Evaluate the Efficacy and Safety of Bevacizumab in Combination With Capecitabine (Xeloda) in Frail Patients With Untreated Metastatic Colorectal Cancer
Brief Title: Bevacizumab Plus Capecitabine (Xeloda) in Patients With Untreated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Oncology Research International (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TORI GI-04; NCT00217685 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab Plus Capecitabine (Experimental): Bevacizumab 7.5 mg/kg every 3 weeks will be administered interavenously (IV) to the enrolled patients. Oral capecitabine 1000 mg/m^2 twice daily for 14 days followed by 7 days off every 21 days. Treatment will continue until disease progression, unacceptable toxicity, or withdrawal of patient consent.
  Interventions: Drug: Capecitabine (Xeloda); Drug: Bevacizumab

INTERVENTIONS:
Drug: Capecitabine (Xeloda) — 1000mg/m^2 administered orally twice daily for two weeks followed by one week rest period
Drug: Bevacizumab — 7.5 mg/kg IV will be administered every 3 weeks

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the bevacizumab and capecitabine combination in frail patients with untreated metastatic colorectal cancer.

DETAILED DESCRIPTION:
The study will evaluate the tolerability, safety, and feasibility of combination bevacizumab and capecitabine in a small number of frail patients with metastatic colorectal cancer who have a compromised performance status. Preclinical studies suggest that the combination of chemotherapy and anti-angiogenic therapy offer an increased anti-tumor effect compared with either treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the colon at first diagnosis
* Stage IV disease, with at least one measurable lesion according to the RECIST criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 2
* No prior chemotherapy for metastatic colorectal cancer
* Prior adjuvant chemotherapy is permitted.
* At least 28 days since prior surgery
* If female of childbearing potential, pregnancy test is negative and willing to use effective contraception while on treatment and for at least 3 months thereafter.
* Required laboratory values:

  * Absolute neutrophil count > 1.5 x 10^9/L
  * Hemoglobin > 9.0 g/dL
  * Platelet count > 100 x 10^9/L
  * Creatinine < 2.0 mg/dL
  * Total bilirubin < 1.5 x upper limit of normal (ULN) (Patients with documented Gilbert's syndrome are eligible.)
  * Alkaline phosphatase and AST/ALT within the following parameters. In determining eligibility, the more abnormal of the two values (AST or ALT) should be used:

    * Alkaline phosphate and AST/ALT < or = ULN
    * Alkaline phosphate > 1x but < or = 2.5x and AST/ALT < or = ULN
    * Alkaline phosphate > 2.5x but < or = 5x and AST/ALT < or = ULN
    * Alkaline phosphate < or = ULN and AST/ALT > 1x but < or = 1.5x
    * Alkaline phosphate > 1x but < or = 2.5 x and AST/ALT > 1x but < or = 1.5x
    * Alkaline phosphate < or = ULN and AST/ALT > 1x but < or = 2.5x

Exclusion Criteria:

* Prior chemotherapy for metastatic colorectal cancer
* Prior treatment with an anti-angiogenic agent
* Concurrent therapy with any other non-protocol anti-cancer therapy
* Current or prior history of central nervous system or brain metastases
* Presence of neuropathy > grade 2 (NCI-Common Toxicity Criteria (CTC) version 3.0) at baseline
* Presence of any non-healing wound, fracture, or ulcer, or the presence of clinically significant (> grade 2) peripheral vascular disease
* History of any other malignancy within the past 5 years, with the exception of non-melanoma skin cancer or carcinoma-in-situ of the cervix
* Clinically significant cardiovascular disease (e.g., blood pressure [BP] > 150/100, myocardial infarction or stroke within the past 6 months, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Active peptic ulcer disease, inflammatory bowel disease, or other gastrointestinal condition increasing the risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning therapy
* Active infection requiring parenteral antimicrobials
* The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of the drugs in this protocol or place the subject at undue risk for treatment complications
* Inability to comply with the study protocol or follow-up procedures
* Pregnancy or lactation
* A history of a severe hypersensitivity reaction to bevacizumab, or capecitabine or other drugs formulated with polysorbate 80.
* Evidence of bleeding diathesis or coagulopathy.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of the need for a major surgical procedure during the course of the study; minor surgical procedure, fine needle aspiration or core biopsy within 7 days prior to Day 0
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Unstable angina
* Urine protein creatinine ratio greater than or equal to 1.
* Therapeutic anticoagulation with oral anticoagulation medications, specifically coumarins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arash Naeim, MD, PhD, Study Chair — University of California, Los Angeles; Randy Hecht, MD, Study Chair — University of California, Los Angeles
Locations (12):
- United States (12):
  - Central Hematology Oncology Medical Group, Inc., Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Virginia K. Crosson Cancer Center, Fullerton, California
  - Pacific Shores Medical Group, Long Beach, California
  - UCLA Medical Center, Los Angeles, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Wilshire Oncology Medical Group, Inc., Pomona, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: October 2005 to February 2009 Types of location: Academic medical oncology clinical and community medical oncology clinics
Groups:
- Bevacizumab Plus Capecitabine: Bevacizumab 7.5 mg/kg every 3 weeks will be administered interavenously (IV) to the enrolled patients. Oral capecitabine 1000 mg/m^2 twice daily for 14 days followed by 7 days off every 21 days. Treatment will continue until disease progression, unacceptable toxicity, or withdrawal of patient consent.
  Capecitabine (Xeloda): 1000mg/m2 administered orally twice daily for two weeks followed by one week rest period
  Bevacizumab: 7.5 mg/kg IV will be administered every 3 weeks
Period: Treatment Period
Arm/Group | Bevacizumab Plus Capecitabine
Started | 45
Completed | 45
Not Completed | 0
Period: Follow-up
Arm/Group | Bevacizumab Plus Capecitabine
Started | 45
Completed | 41
Not Completed | 4
Not completed — Progressive Disease | 4

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 79 [54 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 36
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 45
Eastern Cooperative Oncology Group (ECOG) [Number; unit: subjects] — ECOG Grade Evaluated by Physical Exam 0 Fully active, able to carry on all predisease activities with restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Out of bed > 50%
  3. Capable of only limited self-care, confined to bed or chair > 50% waking hours
  4. Completely disabled, cannot carry on any self-care, totally confined to bed or chair
  subjects
    Score of 1 | 17
    Score of 2 | 28

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression
Description: Progression Free Survival (PFS)- the interval from the date of enrollment to the first documented date of disease progression, death due to cancer, or the last date of a definitive assessment (not an unknown assessment) at which the patient is known to be progression-free. If there is an unknown assessment, then (a) if the next subsequent definitive assessment is complete response (CR), partial response (PR), or stable disease (SD), the patient is considered to be progression-free at the date of the subsequent definitive assessment and PFS is calculated as above; (b) if the next subsequent definitive assessment is progressive disease (PD), the patient is considered to be a failure at the time of the (earliest) assessment of unknown preceding the documented disease progression (i.e. PFS is back-dated to the date of the unknown assessment) and (c) if there is no subsequent definitive assessment, PFS for the patient is considered to be a censored observation at the date
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab Plus Capecitabine: Bevacizumab 7.5 mg/kg every 3 weeks will be administered intravenously (IV) to the enrolled patients. Oral capecitabine 1000 mg/m^2 twice daily for 14 days followed by 7 days off every 21 days. Treatment will continue until disease progression, unacceptable toxicity, or withdrawal of patient consent.
Arm/Group | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 45
months | 6.87 [5.1 to 11.5]

2. Primary Outcome: Number of Subjects Requiring Dose Modifications
Description: Number of Subjects that required Bevacizumab or Capecitabine dose modifications, delay, reduction or discontinuation due to adverse reactions.
Time Frame: 3 months
Population: all subjects that received chemotherapy
Measure: Number; unit: participants
Arm/Group | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 45
participants
  Delay in Bevacizumab Dose | 15
  Discontinuation of Bevacizumab | 14
  Delay in Capec itabineDose | 8
  Reduction of Capecitabine Dose | 13
  Discontinuation of Capecitabine | 16

3. Secondary Outcome: Response Rates
Description: Evaluation of target lesions Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: every 21 days up to 12 months
Measure: Number; unit: participants
Groups:
- Bevacizumab Plus Capecitabine: Bevacizumab 7.5 mg/kg every 3 weeks will be administered intravenously (IV) to the enrolled patients. Oral capecitabine 1000 mg/m2 twice daily for 14 days followed by 7 days off every 21 days. Treatment will continue until disease progression, unacceptable toxicity, or withdrawal of patient consent.
Arm/Group | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 45
participants
  Complete Response | 2
  Partial Response | 14
  Stable Disease | 16
  Progression | 9
  Not Evaluable | 4

4. Secondary Outcome: Quality of Life of Patients
Description: Functional Assessment of Cancer Therapy-Colorectal (FACT-C) Trial Outcome Index (TOI) - a questionnaire assessing quality of life concerns pertinent to colorectal cancer patients. Questions address Physical, Emotional and Functional Well-Being. Scale: Not at all (0), A little bit (1), Somewhat (2), Quite a bit (3), and very much (4). Higher numbers indicate a better state of well being. Scale 0 -136. Higher numbers indicating a better state of well-being.
  The Overall scores for the FACT-C Composite scale range between 0-100 with higher scores indicating a better state of well being.
  The EQ VAS= Euro Quality of Life 5 Dimension Self Reported Healthstate. It records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labeled 0 'Best imaginable health state' and 100 'Worst imaginable health state'.
Time Frame: Baseline, Cycle 2, and End of Study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 45
score on a scale
  Baseline FACT-C Trial outcome index (TOI) | 62.85 (12.12)
  Cycle 2 FACT-C TOI | 66.31 (10.32)
  End of Study FACT-C TOI | 62.09 (12.12)
  Baseline FACT-C Composite | 99.87 (19.87)
  Cycle 2 FACT-C Composite | 105.38 (17.02)
  End of Study FACT-Composite | 98.61 (21.73)
  Baseline EQ-5D VAS | 61.76 (23.17)
  Cycle 2 EQ-5D VAS | 68.59 (22.26)
  End of Study EQ-5D VAS | 66.54 (23.18)

ADVERSE EVENTS:
Time Frame: From time of consent evaluated every 21 days until 30 days after last treatment, up to 1 year.
Description: Systemic adverse event assessment occurred every through investigator assessment during the Treatment period
Arm/Group | Bevacizumab Plus Capecitabine
Serious Adverse Events (participants affected / at risk) | 45/45
Other Adverse Events (participants affected / at risk) | 30/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Plus Capecitabine (N=45)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Fatigue (General disorders) | 6 (6)
Hand Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 6 (6)
Dehydration (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Mucositis (Gastrointestinal disorders) | 2 (2)
Pain-Abdomen (General disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Cerebral vascular accident (Nervous system disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Dyspepsia (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage-GI (Gastrointestinal disorders) | 1 (1)
Obstruction (Gastrointestinal disorders) | 2 (2)
Liver Failure (Hepatobiliary disorders) | 1 (1)
Renal Failure (Hepatobiliary disorders) | 1 (1)
Infarction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Plus Capecitabine (N=45)
Fatigue (General disorders) | 30 (30)
Diarrhea (Gastrointestinal disorders) | 28 (28)
Hand Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 24 (24)
Nausea (Gastrointestinal disorders) | 21 (21)
Mucositis (Gastrointestinal disorders) | 16 (16)
Anorexia (Gastrointestinal disorders) | 15 (15)
Anemia (Blood and lymphatic system disorders) | 13 (13)
Neuropathy (Nervous system disorders) | 11 (11)
Pain-Abdomen (Nervous system disorders) | 10 (10)
Hypertension (Vascular disorders) | 10 (10)
Vomiting (Gastrointestinal disorders) | 9 (9)
Dry Skin (Skin and subcutaneous tissue disorders) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Leukopenia (Blood and lymphatic system disorders) | 7 (7)
Proteinuria (Renal and urinary disorders) | 7 (7)
Dehydration (Gastrointestinal disorders) | 7 (7)
Hemorrhage-Nose (Blood and lymphatic system disorders) | 6 (6)
Weight Loss (Metabolism and nutrition disorders) | 5 (5)
Pain-Head (Nervous system disorders) | 5 (5)
Memory Impairment (General disorders) | 5 (5)
Dizziness (Ear and labyrinth disorders) | 5 (5)
Edema-limb (Blood and lymphatic system disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
This was a small study with only 45 participants who received study treatment. With such a small sample size the study does not have the statistical power to make categorical assessments or statements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No